CLINICAL TRIAL: NCT07294274
Title: Construction and Clinical Validation Study of a Prediction Model for Depression After Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Min Su (Other)
Collaborators: Chongqing Traditional Chinese Medicine Hospital (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 20251114
Record Dates: First submitted 2025-11-27; First posted 2025-12-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group of PSD: The patient was diagnosed with PSD.
  Interventions: Diagnostic Test: Group patients based on whether they have been diagnosed with PSD.
- NPSD: The patient was not diagnosed with PSD.
  Interventions: Diagnostic Test: Group patients based on whether they have been diagnosed with PSD.

INTERVENTIONS:
Diagnostic Test: Group patients based on whether they have been diagnosed with PSD. — Group patients based on whether they have been diagnosed with PSD.

SUMMARY:
Post-stroke depression (PSD) is the most common neuropsychiatric disorder after a stroke, with an incidence rate of 20% to 60%. PSD is not only associated with higher mortality rates, poorer recovery, more obvious cognitive impairments, greater economic burdens, and lower quality of life, but also brings additional medical expenses and care pressure to families. Society also needs to bear higher medical costs. Currently, the early diagnosis of PSD is difficult, which may lead to poor prognosis after stroke. This study aims to utilize machine learning technology to integrate multi-dimensional indicators of patients with ischemic stroke, establish a risk prediction model for PSD, and assist in early, accurate, and individualized assessment of PSD risk in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke;
* Admission within 7 days of symptom onset;
* The patient and/or the family members sign a written informed consent form.

Exclusion Criteria:

* Confusion of consciousness,severe cognitive impairment, etc
* Individuals with a history of depression, schizophrenia, bipolar disorder, etc;
* Individuals unable to participate in neuropsychological examinations due to hearing im pairments, lack of coordination, or neurological deficits, including se vere aphasia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute ischemic stroke patients who may develop post-stroke depression
Sampling Method: Non-Probability Sample
Enrollment: 488 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
The number of post-stroke depression (PSD) that occurs 3 months after stroke | 3 months after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China